CLINICAL TRIAL: NCT05589779
Title: Relationship Between Cardiovascular Disease in Asthma and Eosinophil Subtypes and Biomarkers of Bronchial Remodeling.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-ASM-2022-89
Record Dates: First submitted 2022-10-10; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Asthma; Cardiovascular Diseases
Keywords: Asthma; Cardiovascular Diseases; Chronic inflammation; Bronchial remodeling; Eosinophilia
MeSH Terms: conditions — Asthma; Cardiovascular Diseases; Eosinophilia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With cardiovascular disease: Asthma patients with cardiovascular disease
  Interventions: Other: Asthma and cardiovascular disease
- Without cardiovascular disease: Asthma patients without cardiovascular disease
  Interventions: Other: Asthma and cardiovascular disease

INTERVENTIONS:
Other: Asthma and cardiovascular disease — To know the clinical and inflammatory characteristics of patients with asthma and associated cardiovascular disease, as well as their relationship with eosinophil subtypes, biomarkers of chronic inflammation and bronchial remodeling.

SUMMARY:
To know the clinical and inflammatory characteristics of patients with asthma and associated cardiovascular disease.

DETAILED DESCRIPTION:
Recent studies have shown that asthma could be a risk factor for cardiovascular disease, especially in the female and late-onset subgroups. The two entities share several risk factors, such as chronic inflammation and bronchial remodeling. Eosinophilia, characteristic of asthma, has also been described as a predictor of cardiovascular mortality.

The aim of this study is to determine the clinical and inflammatory characteristics of patients with asthma and associated cardiovascular disease, as well as their relationship with eosinophil subtypes, biomarkers of chronic inflammation and bronchial remodeling.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of asthma
* Signed informed consent

Exclusion Criteria:

* Age under 18 years old
* Age over 99 years old
* Pneumological diseases other than asthma
* Active oncological diseases or with end of treatment <5 years
* Autoimmune or systemic inflammatory diseases

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthmatic patients with and without cardiovascular disease
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Clinical characteristics of patients with asthma | 1 year
  Spirometry with bronchodilator testing
Associated cardiovascular disease type | 1 year
  Cardiac infarction, stroke or peripheral artery disease

SECONDARY OUTCOMES:
Eosinophil subtypes | 1 year
  Eosinophil subtypes of patients with asthma and cardiovascular disease
Biomarkers of chronic inflammation | 1 year
  Transforming growth factor-β, interleukin-5, interleukin-13, interleukin-25 and interleukin-3
Bronchial remodeling | 1 year
  Bronchial remodeling of patients with asthma and cardiovascular disease measured by analysis of images obtained by thoracic CT scanning

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Result] Zhang B, Li ZF, An ZY, Zhang L, Wang JY, Hao MD, Jin YJ, Li D, Song AJ, Ren Q, Chen WB. Association Between Asthma and All-Cause Mortality and Cardiovascular Disease Morbidity and Mortality: A Meta-Analysis of Cohort Studies. Front Cardiovasc Med. 2022 Mar 17;9:861798. doi: 10.3389/fcvm.2022.861798. eCollection 2022. PMID 35369308
- [Result] Wang L, Gao S, Yu M, Sheng Z, Tan W. Association of asthma with coronary heart disease: A meta analysis of 11 trials. PLoS One. 2017 Jun 13;12(6):e0179335. doi: 10.1371/journal.pone.0179335. eCollection 2017. PMID 28609456
- [Result] Xu M, Xu J, Yang X. Asthma and risk of cardiovascular disease or all-cause mortality: a meta-analysis. Ann Saudi Med. 2017 Mar-Apr;37(2):99-105. doi: 10.5144/0256-4947.2017.99. PMID 28377538
- [Result] Liu H, Fu Y, Wang K. Asthma and risk of coronary heart disease: A meta-analysis of cohort studies. Ann Allergy Asthma Immunol. 2017 Jun;118(6):689-695. doi: 10.1016/j.anai.2017.03.012. Epub 2017 Apr 19. PMID 28433577
- [Result] Guite HF, Dundas R, Burney PG. Risk factors for death from asthma, chronic obstructive pulmonary disease, and cardiovascular disease after a hospital admission for asthma. Thorax. 1999 Apr;54(4):301-7. doi: 10.1136/thx.54.4.301. PMID 10092690
- [Result] Banno A, Reddy AT, Lakshmi SP, Reddy RC. Bidirectional interaction of airway epithelial remodeling and inflammation in asthma. Clin Sci (Lond). 2020 May 15;134(9):1063-1079. doi: 10.1042/CS20191309. PMID 32369100
- [Result] Lee HM, Liu MA, Barrett-Connor E, Wong ND. Association of lung function with coronary heart disease and cardiovascular disease outcomes in elderly: the Rancho Bernardo study. Respir Med. 2014 Dec;108(12):1779-85. doi: 10.1016/j.rmed.2014.09.016. Epub 2014 Oct 6. PMID 25448311
- [Result] Kannel WB, Hubert H, Lew EA. Vital capacity as a predictor of cardiovascular disease: the Framingham study. Am Heart J. 1983 Feb;105(2):311-5. doi: 10.1016/0002-8703(83)90532-x. No abstract available. PMID 6823813
- [Result] Schroeder EB, Welch VL, Couper D, Nieto FJ, Liao D, Rosamond WD, Heiss G. Lung function and incident coronary heart disease: the Atherosclerosis Risk in Communities Study. Am J Epidemiol. 2003 Dec 15;158(12):1171-81. doi: 10.1093/aje/kwg276. PMID 14652302
- [Result] Sin DD, Wu L, Man SF. The relationship between reduced lung function and cardiovascular mortality: a population-based study and a systematic review of the literature. Chest. 2005 Jun;127(6):1952-9. doi: 10.1378/chest.127.6.1952. PMID 15947307
- [Result] Rothenberg ME, Hogan SP. The eosinophil. Annu Rev Immunol. 2006;24:147-74. doi: 10.1146/annurev.immunol.24.021605.090720. PMID 16551246
- [Result] Januskevicius A, Jurkeviciute E, Janulaityte I, Kalinauskaite-Zukauske V, Miliauskas S, Malakauskas K. Blood Eosinophils Subtypes and Their Survivability in Asthma Patients. Cells. 2020 May 18;9(5):1248. doi: 10.3390/cells9051248. PMID 32443594
- [Result] Mesnil C, Raulier S, Paulissen G, Xiao X, Birrell MA, Pirottin D, Janss T, Starkl P, Ramery E, Henket M, Schleich FN, Radermecker M, Thielemans K, Gillet L, Thiry M, Belvisi MG, Louis R, Desmet C, Marichal T, Bureau F. Lung-resident eosinophils represent a distinct regulatory eosinophil subset. J Clin Invest. 2016 Sep 1;126(9):3279-95. doi: 10.1172/JCI85664. Epub 2016 Aug 22. PMID 27548519